CLINICAL TRIAL: NCT06517212
Title: Adjuvant Tirzepatide Plus Standard of Care Endocrine Therapy in Patients With Obesity or Overweight Who Have Hormone Receptor-positive, HER2-negative, Node-positive Early Breast Cancer, With Molecular Residual Disease (MRD), as Determined by Circulating Tumor DNA (ctDNA)
Brief Title: Tirzepatide Weight Loss for MRD+ Early Breast Cancer
Acronym: TRIM-EBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 024-273
Record Dates: First submitted 2024-07-02; First posted 2024-07-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Cancers
Keywords: TRIM; TRIM EBC; TRIM-EBC; tirzepatide; MRD; ctDNA
MeSH Terms: conditions — Breast Neoplasms | interventions — Tirzepatide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- tirzepatide (Experimental): Patients will be treated with tirzepatide 15mg subcutaneously (SC) weekly (starting with 2.5mg SC weekly and increasing by 2.5mg monthly over 6 months) and will be monitored closely for tolerability, safety, and weight loss. Patients may be treated with tirzepatide for up to 2 years on trial if they remain without evidence of metastatic disease recurrence and provided there's demonstrated safety of tirzepatide with associated weight loss.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Patients will receive tirzepatide once weekly for up to 2 years.
  Other Names: ZepBound

SUMMARY:
This trial aims to asses if tirzepatide-induced weight loss will lead to metabolic and hormonal changes in hormone receptor-positive (HR+), human epidermal growth factor receptor-negative (HER2-), node-positive (N+) high risk early breast cancer patients with obesity or overweight, inhibiting the growth and survival of micrometastatic disease and leading to clearance of tumor-informed circulating tumor DNA (ctDNA) and freedom from the development of metastatic disease.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if tirzepatide induced weight loss effects survival outcomes in high risk early breast cancer patients. The main questions it aims to answer are:

1. Does tirzepatide-induced weight loss lead to clearance of plasma ctDNA in the adjuvant setting in patients with obesity or overweight who have HR+, HER2-, N+ early breast cancer who are at high risk of recurrence, and
2. Does tirzepatide-induced weight loss prevent the development of overt metastatic disease and improve distant disease-free survival, in the two-year period following first detection of ctDNA in patients with obesity or overweight who have HR+, HER2-, N+ early breast cancer who are at high risk of recurrence.

Researchers will assess clinical outcomes after the first 20 patients are enrolled and have taken tirzepatide for at least 6 months. If at least three of the first 20 evaluable patients demonstrate clearance of ctDNA on tirzepatide, or at least ten of the first 20 patients remain alive and free of distant metastatic disease during the two-year period following initial detection of ctDNA using the Kaplan-Meier method, an additional 28 ctDNA-positive patients will be enrolled.

Patients will screen for ctDNA every 3 months for up to 3 years or until ctDNA positivity, whichever comes first. Once positive, they will undergo radiologic imaging to confirm the absence of frank metastatic disease. If confirmed, patients will receive tirzepatide once weekly for up to 2 years, visit the clinic monthly for the first 6 months, and every other month thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients ≥18 years of age
2. Have a diagnosis of node-positive, hormone receptor-positive (ER+ > 10%), and HER2-negative breast cancer within the past 15 years per the American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines

   1. If patients have synchronous bilateral ER+ breast cancers, tissue from both primary cancers should be submitted for next-generation sequencing (NGS) to inform ctDNA testing
   2. Patients with multifocal/multicentric cancers are eligible and the largest focus of cancer should be submitted for NGS evaluation. If tested, all tumor foci must meet have ER > 10%
   3. For patients who received neoadjuvant therapy and have discordant hormone receptor and/or HER2 results between the diagnostic biopsy (pre-treatment) and the surgical pathology (post-neoadjuvant treatment), the hormone receptor status and HER2 status of the post-treatment specimen will determine eligibility
3. Overweight or obesity defined as body mass index (BMI) > 27 kg/m2
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
5. Have received at least 1 year of or having completed standard neo/adjuvant endocrine therapy. If adjuvant cyclin dependent kinase (CDK) 4/6 inhibitor therapy was prescribed, patients must have completed this therapy
6. Positive ctDNA blood test as determined by the Haystack Oncology Haystack MRD tumor-informed ctDNA assay
7. Patients must have formalin-fixed paraffin-embedded (FFPE) tissue from the primary tumor available for submission to Haystack Oncology to perform whole genome sequencing (WGS) to build customized mutation panel to monitor for plasma ctDNA
8. No clinical evidence of metastatic breast cancer found on history, physical examination, complete blood count (CBC), comprehensive metabolic panel (CMP), and radiologic imaging following a finding of positive ctDNA
9. Have adequate hematologic function, defined by:

   1. Absolute neutrophil count (ANC) >1500/µL
   2. Platelet count ≥100,000/ µL
   3. Hemoglobin ≥9 g/dL or ≥5.6 mmol/L
10. Have adequate liver function, defined by:

    1. Aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤3 x the upper limit of normal (ULN)
    2. Total bilirubin ≤1.5 x ULN OR direct bilirubin ≤ULN for patients with total bilirubin levels >1.5 × ULN
11. Have adequate renal function, defined by:

    a. Serum creatinine ≤1.5 x ULN or calculated creatinine clearance of ≥30 mL/min
12. Patients must be accessible for treatment and follow-up
13. All patients must be able to understand the investigational nature of the study and give written informed consent prior to study entry

Exclusion Criteria:

1. Prior bariatric surgery and/or endoscopic procedures for weight loss (e.g., intragastric balloon, sleeve gastrostomy) following diagnosis of breast cancer
2. Treatment with a GLP-1/Glucagon receptor agonist, GIP/GLP-1/Glucagon receptor agonist, GIP/GLP receptor agonist, or any combinations with GLP-1 receptor agonist therapies within the last 3 months
3. History of severe hypersensitivity reaction to GLP-1/Glucagon receptor agonist, GIP/GLP-1/Glucagon receptor agonist, or any combinations with GLP-1 receptor agonist therapies
4. Insulin-dependent diabetes
5. Has clinical evidence of diabetic retinopathy
6. Clinical evidence or suspicion of metastatic breast cancer
7. Current or past invasive cancers, other than breast cancer, are not allowed except for:

   1. Adequately treated basal or squamous cell carcinoma of the skin
   2. Previously diagnosed invasive cancer treated with curative intent, with no evidence of disease recurrence for at least 5 years, and are considered low risk for future recurrence by the treating physician
8. Patients with a second synchronous primary HER2-positive or triple negative breast cancer
9. Has an active infection requiring systemic therapy
10. Has a known history of human immunodeficiency virus (HIV) or active or persistent hepatitis B or hepatitis C virus
11. Has significant cardiovascular disease, such as:

    1. History of stroke, myocardial infarction, acute coronary syndrome, or coronary angioplasty/stenting/bypass grafting within the last 6 months
    2. Congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV, or history of CHF NYHA class III or IV.
12. Has a known history of active tuberculosis
13. Women who are pregnant or lactating. All patients of reproductive potential must agree to use effective contraception from time of study entry until at least 3 months after the last administration of study drug
14. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation such as:

    1. severe impaired lung functions as defined as spirometry and diffusing capacity of lung for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
    2. liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C)
    3. history of gastroparesis, impaired gastrointestinal (GI) function, or GI disease that may significantly alter the absorption of the study drug (e.g., ulcerative diseases, uncontrolled nausea vomiting and/or diarrhea, malabsorption syndrome, or small bowel resection)
15. Has a history of pancreatitis or current symptoms of untreated cholelithiasis
16. Has a family history of Multiple Endocrine Neoplasia Syndrome Type 2 (MEN 2) or medullary thyroid cancer (MTC)
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's full participation for the full duration of the study, or results in trial participation not being in the patient's best interest, in the opinion of the Treating Physician
18. Has received an investigational agent within 4 weeks prior to study treatment; investigational monoclonal antibodies should have a 4-week (28 day) or 5 half-life washout period
19. Any other investigational or anti-cancer treatments while participating in this study with the exception of standard adjuvant endocrine therapy, zoledronic acid, or denosumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
ctDNA efficacy | 2 years
  Clearance of the presence of plasma ctDNA within two years of documented ctDNA positivity at time of study entry.
distant disease-free survival efficacy | 2 years
  Percentage of patients alive and free of distant metastatic disease at 2 years following detection of ctDNA at the time of study entry.

SECONDARY OUTCOMES:
ctDNA kinetic changes using Haystack MRD | 2 years
  Differences in ctDNA kinetics between patients who clear ctDNA versus patients who do not clear ctDNA while on tirzepatide using the Haystack MRD assay.
Number of patients with Treatment-Related Adverse Events (Safety and Tolerability) | 2 years
  Number of patients with treatment related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
weight loss | 2 years
  Percentage of weight loss observed on tirzepatide associated with clearance or persistence of ctDNA in patients receiving standard adjuvant endocrine therapy.

OTHER OUTCOMES:
time to recurrence | 5 years
  Breast cancer distant disease-free survival, defined as the time from beginning tirzepatide therapy to the time of distant disease recurrence or death, over five years in ctDNA-positive patients who clear ctDNA versus patients who do not clear ctDNA while on tirzepatide.
exploratory molecular changes via Next Generation Sequencing (NGS), Flow Cytometry, and Reverse Phase Protein Array (RPPA) | 5 years
  Exploratory analysis of metabolic, hormonal and immune cell changes associated with weight loss on tirzepatide in early breast cancer patients. Exploratory analyses may include NGS, Flow Cytometry, and RPPA.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce A O'Shaughnessy, MD, Principal Investigator — Baylor Scott and White Research Institute
Locations (1):
- Baylor University Medical Center, Baylor Charles A Sammons Cancer Center, Dallas, Texas, United States